CLINICAL TRIAL: NCT05463263
Title: An Open-Label, First in Human, Phase 1/2 to Evaluate Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of the CTPS1 Inhibitor STP938 In Adult Subjects With Relapsed/Refractory B-Cell and T-Cell Lymphomas
Brief Title: A Phase 1/2 Study of STP938 for Adult Subjects With Relapsed/Refractory B-Cell and T-Cell Lymphomas
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Step Pharma, SAS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STP938-101
Record Dates: First submitted 2022-06-30; First posted 2022-07-18 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-12

CONDITIONS: Lymphoma, B-Cell; Lymphoma, T-Cell
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, T-Cell

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to a dose level of STP938 (Phase 1) or an expansion cohort (Phase 2) at the time of their enrollment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Part 1, Dose Escalation) (Experimental): Up to 5 dose levels with STP938 administered as oral monotherapy
  Interventions: Drug: STP938
- Phase 2 (Part 2; expansion) (Experimental): At defined dose level(s) with STP938 administered as oral monotherapy
  Interventions: Drug: STP938

INTERVENTIONS:
Drug: STP938 — Small molecule

SUMMARY:
The Phase 1 part of the study is a dose escalation of STP938 as monotherapy.

The Phase 2 part of the study is cohort expansion of STP938 as a monotherapy in 5 different B and T cell lymphomas.

DETAILED DESCRIPTION:
The drug STP938 is an inhibitor of an enzyme called cytidine triphosphate synthase 1 (CTPS1). CTPS1, and a very similar enzyme cytidine triphosphate synthase 2 (CTPS2), control the final step in the production of the cytidine triphosphate (CTP). CTP is an essential building block of deoxyribonucleic acid (DNA) and ribonucleic acid (RNA). Studies of people with inherited mutations of the CTPS1 gene indicate that certain types of blood cells required CTPS1 in order to divide rapidly, whereas other cells in the body use the CTPS2 enzyme. Based on these observations, it is expected that blocking CTPS1, using the drug STP938, may be an effective treatment for certain types of cancer that arise from blood cells.

The purpose of this study is to see if STP938 is effective at treating different types of lymphoma. STP938 will be given as a tablet. Blood samples will be taken during the study in order to understand the effects of STP938 on the lymphoma and on the rest of the body. The main outcome of the first part of the study is to see if STP938 can be given safely to patients with lymphoma, and to work out the best dose of STP938. The main outcome of the second part of the study is to see if ST938 is effective in treating different types of lymphoma.

ELIGIBILITY:
Main Inclusion Criteria:

* Signed and dated informed consent, and able to comply with the study procedures and any locally required authorization.
* Male or female aged ≥ 18 years.
* Relapsed/refractory patients with histologically confirmed diagnosis of B cell or T cell lymphoma
* Must have received at least 2 prior systemic therapies and have no treatment options known to provide clinical benefit
* Must have measurable disease per Lugano lymphoma classification except for cutaneous T-cell lymphoma (CTCL) which is measured via International Society for Cutaneous Lymphomas (ISCL)/ European Organization of Research and Treatment of Cancer (EORTC).
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Life expectancy > 3 months as assessed by the Investigator.
* Adequate organ function (bone marrow, hepatic, renal function and coagulation).
* All toxicities (except alopecia) from prior cancer treatments or procedures must have resolved to ≤Grade 1 or returned to baseline levels prior to enrollment.

Main Exclusion Criteria:

* Pregnant or breastfeeding females and women of child bearing potential or males unwilling to comply with contraception requirements.
* Known carcinomatous meningitis or central nervous system (CNS) involvement with lymphoma.
* Active malignancy within 2 years of study enrollment
* Prior radiation or surgical resection of their lymphoma without additional sites of measurable disease outside of the radiation field or subjects who have received prior radiation or surgical resection of their lymphoma ≤2 weeks prior to the first dose of study drug.
* Systemic cancer treatments, monoclonal antibody-directed therapies, other investigational agents within 4 weeks before enrollment, or <5 half-lives since completion of previous investigational therapy, whichever is shorter.
* Uncontrolled intercurrent illness.
* Immunocompromised subjects with increased risk of opportunistic infections or history of opportunistic infection in the last 12 months.
* Known active or chronic hepatitis B or active hepatitis C virus (HCV) infection.
* Subjects who have received a live vaccine within 30 days prior to study enrollment or whilst participating in the study.
* Subjects with corrected QT interval >470 msec based on averaged triplicate electrocardiogram (ECG) readings at the Screening Visit using the QT interval corrected for heart rate using Fridericia's method (QTcF).
* Subjects who received a severe acute respiratory syndrome coronavirus 2 vaccine ≤3 weeks prior to study drug dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability (Phase 1 / Dose Escalation) | Through study completion, an average of 9 months
  Incidence of dose limiting toxicities (DLTs), serious adverse events (SAEs), treatment-emergent adverse events (TEAEs)
Objective Response Rate (ORR) (Phase 2 / Dose Expansion) | Through study completion, an average of 9 months
  ORR is defined as the proportion of subjects achieving a confirmed response (complete response [CR] or partial response [PR]). Evaluation of ORR will be via standard response criteria

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of STP938 including effects of food on absorption (Phase 1 / Dose Escalation) | 16 Days
  Pharmacokinetic parameter from plasma STP938 levels
Time to reach maximum concentration (TMax) of STP938 including effects of food on absorption (Phase 1 / Dose Escalation) | 16 Days
  Pharmacokinetic parameter from plasma STP938 levels
Area under the curve (AUC) of STP938 including effects of food on absorption (Phase 1 / Dose Escalation) | 16 Days
  Pharmacokinetic parameter from plasma STP938 levels
Evaluate preliminary clinical activity of STP938 (Phase 1) | Through study completion, an average of 9 months
  Evaluation of ORR using standard response criteria
Evaluate best overall response of STP938 (Phase 1 / Phase 2) | Through study completion, an average of 9 months
  Evaluation of best overall response (Complete response [CR], Partial response [PR], Stable disease [SD], Progression of disease [PD], Not evaluable, Not applicable) using standard response criteria
Evaluation Time To Respond (Phase 1 / Phase 2) | Through study completion, an average of 9 months
  Time to response (TTR) defined as the time from first dose of STP938 to the date of first CR or PR response assessment
Evaluation Duration of Response (Phase 1 / Phase 2) | Through study completion, an average of 9 months
  Duration of response (DoR) is defined as the time, in days, from the date measurement criteria that are first met for CR or PR (whichever is first recorded) to the first date that relapse, progressive disease or death, whichever occurs first
Evaluation Progression Free Survival (Phase 1 / Phase 2) | Through study completion, an average of 9 months
  Progression-free survival (PFS) is defined as the time from first STP938 dose to the date of disease progression or death, whichever occurs first
Evaluation of Complete Response Rate (Phase 2) | Through study completion, an average of 9 months
  Complete Response Rate using standard response criteria
Safety and Tolerability (Phase 2 / Dose Expansion) | Through study completion, an average of 9 months
  Incidence of SAEs and TEAEs

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Higgins, Study Director — Step Pharma
Locations (15):
- United States (3):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Memorial Sloan Kettering, New York, New York
- France (5):
  - The Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHU de Nantes, Nantes
  - Hôpital Saint-Louis, Paris
  - Institut Gustave Roussy, Villejuif
- United Kingdom (7):
  - University Hospitals of Leicester NHS Trust, Leicester
  - Imperial College / Clinical Trials Unit, Hammersmith Hospital, London
  - The Christie, Manchester
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - The Royal Marsden, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Asnagli H, Minet N, Pfeiffer C, Hoeben E, Lane R, Laughton D, Birch L, Jones G, Novak A, Parker AE, Ludwig H, Fischer A, Latour S, Beer PA. CTP Synthase 1 Is a Novel Therapeutic Target in Lymphoma. Hemasphere. 2023 Mar 28;7(4):e864. doi: 10.1097/HS9.0000000000000864. eCollection 2023 Apr. PMID 37008165